CLINICAL TRIAL: NCT05792228
Title: A Standardized Intervention to Improve the Management of Chemotherapy-induced Nausea and Vomiting in Patients With Head and Neck Squamous Cell Carcinomas
Brief Title: A Standardized Intervention to Improve the Management of Chemotherapy-induced Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ZC20009
Record Dates: First submitted 2023-03-13; First posted 2023-03-31 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Chemotherapy Induced Nausea and Vomiting
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Vomiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group will receive evidence-based, nurse-led standardized management of CINV, including nurse-led risk assessment, education on prevention and control of CINV, antiemetics following guidelines, dietary strategies, relaxation therapy, and follow up.
  Interventions: Other: nurse-led standardized intervention
- The control group (No Intervention): The control group will receive the routine CINV management. Patients are given drugs to prevent and control emesis according to the physicians' individual prescriptions. Nurses provide related education about nausea and vomiting control and recommend patients to drink more water and eat light food. Patients will be given Metoclopramide when they are vomiting.

INTERVENTIONS:
Other: nurse-led standardized intervention — Once the patient in the intervention group decided to undergo cisplatin-based chemotherapy, the nurses would assess the risk factors associated with chemotherapy-induced nausea and vomiting (CINV) and reported to the physicians. During the chemotherapy, nurses would provide education on prevention and control of CINV using web-based approaches. All patients received standard antiemetic regimen, which included Aprepitant, 5-Hydroxytryptamine3-receptor antagonists, and Dexamethasone. If the physician's prescription was not accordance with the standard antiemetic regimen, nurse would remind the physician to adjust the prescription. Patients were recommended to eat small and frequent meals slowly. Overly spicy, fatty, and sweet foods should be avoided. Music relaxation therapy was performed for 60 min each time, once a day, and 3 times in the whole chemotherapy cycle. Follow-up was delivered until the 5th day after chemotherapy.
  Arms: The intervention group

SUMMARY:
The goal of this clinical trial is to investigate the effect of a nurse-led standardized intervention on chemotherapy induced nausea and vomiting (CINV) in patients with head and neck squamous cell carcinoma. The main questions it aims to answer are: (1) what's the best practice to enhance the management of CINV; (2) how's the effect of the nurse-led standardized intervention on CINV in the patients treated with cisplatin-based chemotherapy. Participants in the intervention group will receive evidence-based, nurse-led standardized management of CINV, including nurse-led risk assessment, education on prevention and control of CINV, antiemetics following guidelines, dietary strategies, relaxation therapy, and follow up. Participants in the control group will receive routine care of CINV. The incidence and occurrence degree of CINV and its influence on patients' quality of life will be compared between the two groups.

DETAILED DESCRIPTION:
Chemotherapy with cisplatin is one of the most common treatments for patients with HNSCC, which could very possibly cause severe nausea and vomiting in last up to 5 days after administration of the drug. Nurses play an important role in managing CINV. The goal of this clinical trial is to investigate the effect of a nurse-led standardized intervention on chemotherapy induced nausea and vomiting (CINV) in patients with head and neck squamous cell carcinoma. The main questions it aims to answer are: (1) what's the best practice to enhance the management of CINV; (2) how's the effect of the nurse-led standardized intervention on CINV in the patients treated with cisplatin-based chemotherapy. Best practice to optimize CINV management for HNSCC patients who receive cisplatin-based chemotherapy have been instituted based on evidence. Participants in the intervention group will receive the evidence-based, nurse-led standardized management of CINV. Once the patient in the intervention group decide to undergo cisplatin-based chemotherapy, the nurses would assess the risk factors associated with chemotherapy-induced nausea and vomiting (CINV) and report to the physicians. During the chemotherapy, nurses will provide education on prevention and control of CINV using web-based approaches. All patients will receive standard antiemetic regimen, which includes Aprepitant, 5-HT3 RA, and Dexamethasone. If the physician's prescription are not accordance with the standard antiemetic regimen, nurse would remind the physician to adjust the prescription. Patients will be recommended to eat small and frequent meals slowly. Overly spicy, fatty, and sweet foods should be avoided. Music relaxation therapy will be performed for 60 min each time, once a day, and 3 times in the whole chemotherapy cycle. Follow-up will be delivered until the 5th day after chemotherapy. Guides on how to relieve nausea and vomiting will also be provided. Participants in the control group will receive routine care of CINV. Patients will be given drugs to prevent and control emesis according to the physicians' individual prescriptions. Nurses provide education about nausea and vomiting control and recommend patients to drink more water and eat light food. Patients will be given Metoclopramide when they are vomiting. The incidence and occurrence degree of CINV and its influence on patients' quality of life will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with head and neck squamous cell carcinoma
* receive first cycle of chemotherapy
* receive cisplatin-based chemotherapy
* able to read and write.

Exclusion Criteria:

* experience nausea or vomiting in 24 hours before receiving chemotherapy
* mental disturbance
* disturbance of consciousness
* history of stomach disease or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
The incidence of chemotherapy-induced nausea and vomiting | Five days after administration of cisplatin
  The number of patients who have chemotherapy-induced nausea and vomiting during the first cycle of chemotherapy will be collected.
The degree of chemotherapy-induced nausea and vomiting | Five days after administration of cisplatin
  The degree of chemotherapy-induced nausea and vomiting would be assessed by the Common Terminology Criteria for Adverse Events v3.0 during the first cycle of chemotherapy
The influence of chemotherapy-induced nausea and vomiting on patients' quality of life | Five days after administration of cisplatin
  The influence of chemotherapy-induced nausea and vomiting on patients' quality of life would be assessed by the Functional Living Index-Emesis during the first cycle of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical universtiy cancer institute and hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Cao J, Chen C, Wang Y, Liu M, Han X, Li H. A nurse-led multidomain intervention to improve the management of chemotherapy-induced nausea and vomiting in patients with head and neck cancers: A randomized controlled trial. Eur J Oncol Nurs. 2024 Jun;70:102615. doi: 10.1016/j.ejon.2024.102615. Epub 2024 May 20. PMID 38797114